CLINICAL TRIAL: NCT02750514
Title: A Phase 2, Fast Real Time Assessment of Combination Therapies in Immuno-Oncology Study in Subjects With Advanced Non-Small Cell Lung Cancer (FRACTION-Lung)
Brief Title: An Investigational Immuno-therapy Study to Test Combination Treatments in Patients With Advanced Non-Small Cell Lung Cancer
Acronym: FRACTION-Lung
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The standard of care for the patient population changed and we were unable to accrue any longer.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA018-001
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab; Dasatinib; relatlimab; Ipilimumab; linrodostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Nivolumab (Active Comparator): Nivolumab Monotherapy - Arm associated with this intervention is closed. Nivolumab is no longer given as an active comparator
  Interventions: Biological: Nivolumab
- Nivolumab & Dasatinib (Experimental): Nivolumab in combination with Dasatinib
  Interventions: Biological: Nivolumab; Drug: Dasatinib
- Nivolumab & Relatlimab (Experimental): Nivolumab in combination with Relatlimab
  Interventions: Biological: Nivolumab; Biological: Relatlimab
- Nivolumab & Ipilimumab (Experimental): Nivolumab in combination with Ipilimumab
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab & BMS-986205 (Experimental): Nivolumab in combination with BMS- 986205
  Interventions: Biological: Nivolumab; Drug: BMS-986205

INTERVENTIONS:
Biological: Nivolumab — Arm associated with this intervention is closed. Nivolumab is no longer given as an active comparator.
  Other Names: BMS-936558; MDX-1106; OPDIVO
Drug: Dasatinib
  Other Names: BMS-354825; SPRYCEL
  Arms: Nivolumab & Dasatinib
Biological: Relatlimab
  Other Names: BMS-986016
  Arms: Nivolumab & Relatlimab
Biological: Ipilimumab
  Other Names: BMS-734016; Yervoy
  Arms: Nivolumab & Ipilimumab
Drug: BMS-986205 — Specified dose on specified days
  Arms: Nivolumab & BMS-986205

SUMMARY:
The purpose of this study is to determine whether Nivolumab, in combination with other therapies, is effective in patients with advanced Non-Small Cell lung cancer

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Advanced Non Small Cell Lung Cancer (NSCLC)
* Eastern Cooperative Oncology Group (ECOG) Performance status of ≤ 1
* Life expectancy of at least 3 months from most recent chemotherapy or immunotherapy treatment
* Must have at least 1 lesion with measurable disease

Exclusion Criteria:

* Subjects with certain mutations that have not been treated with a targeted therapy prior to enrollment
* Subjects who need daily oxygen therapy
* People with autoimmune disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (48):
- United States (35):
  - City of Hope National Medical Center, Duarte, California
  - University of Southern California (USC), Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Californa, Los Angeles (UCLA), Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California San Diego, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Maryland - Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber/Harvard Cancer Center, Boston, Massachusetts
  - University of Michigan Health System (UMHS) - University Hospital (University of Michigan Medical Ce, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, The Center for Advanced Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Univ of NC Shool of Medicine, Chapel Hill, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Northwest Cancer Specialists, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The West Clinic, P.C. d/b/a West Cancer Center, Germantown, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Sammons Cancer Center (Uso), Dallas, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Us Oncology, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Washington-Seattle Cancer Care Alliance, Seattle, Washington
- Local Institution, Clayton, Victoria, Australia
- Local Institution, Salzburg, Austria
- Canada (3):
  - Juravinski Cancer Centre, Hamilton Health Sciences-Mcmaster Univeristy's Faculty Of Health Sciences, Hamilton, Ontario
  - University Of Ottawa - The Ottawa Hospital Cancer centre, Ottawa, Ontario
  - Local Institution, Edmonton
- France (3):
  - Local Institution, Paris
  - Local Institution, Toulouse
  - Local Institution, Villejuif
- Italy (2):
  - Local Institution, Milan
  - Local Institution, Rozzano
- Spain (2):
  - Local Institution, Madrid
  - Local Institution, Pamplona
- Local Institution, Lausanne, Switzerland

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total number of participants randomized and treated is 295. Each participant was assigned to 1 of 5 non-consecutive Tracks (based on previous therapy exposure and/or PD-1/PD-L1 expression).
  14 of the 295 participants, after receiving initial treatment, were re-randomized to a second, different treatment (either under a different Track or within the same Track).
Groups:
- Nivolumab: Nivolumab monotherapy 240 mg Q2W administered until completion of 6 cycles (1 cycle=4 weeks)
- Nivolumab + Dasatinib: Nivolumab 240 mg Q2W + Dasatinib 100 mg QD, administered until completion of 6 cycles (1 cycle=4 weeks)
- Nivolumab + BMS986016: Nivolumab 240 mg Q2W + BMS986016 20 mg Q2W, administered until completion of 6 cycles (1 cycle=4 weeks)
- Nivolumab + Ipilimumab: Nivolumab 240 mg Q2W for 12 doses + Ipilimumab 1 mg/kg Q6W for 4 doses, administered until completion of 24 weeks of study
- Nivolumab + BMS986205: Nivolumab 480 mg Q4W + BMS986205 100 mg QD, administered until completion of 6 cycles (1 cycle=4 weeks)
Period: Track 1
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Started | 40 | 4 | 0 | 3 | 0
Completed | 13 (3 participants were re-randomized to track 3 (2 part.) or track 5 (1 part.)) | 2 | 0 | 1 | 0
Not Completed | 27 | 2 | 0 | 2 | 0
Not completed — Disease progression | 20 | 1 | 0 | 1 | 0
Not completed — Adverse event unrelated to study drug | 1 | 0 | 0 | 0 | 0
Not completed — Study drug toxicity | 4 | 1 | 0 | 1 | 0
Not completed — Participant request to discontinue | 1 | 0 | 0 | 0 | 0
Not completed — Other reasons | 1 | 0 | 0 | 0 | 0
Period: Track 2
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Started | 9 | 8 | 2 | 12 | 0
Completed | 3 (2 participants were re-randomized to track 3 (1 part.) or track 5 (1 part.)) | 0 | 0 | 5 (1 participant was re-randomized to track 5) | 0
Not Completed | 6 | 8 | 2 | 7 | 0
Not completed — Disease progression | 4 | 5 | 2 | 5 | 0
Not completed — Adverse event unrelated to study drug | 1 | 0 | 0 | 0 | 0
Not completed — Study drug toxicity | 1 | 2 | 0 | 2 | 0
Not completed — Participant withdrew consent | 0 | 1 | 0 | 0 | 0
Period: Track 3
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Started | 0 | 41 (2 participants had prior treatment in track 1 (1 part.) or track 2 (1 part.)) | 16 (1 participant had prior treatment in track 3) | 18 (5 participants had prior treatment in track 1 (1 part.) or track 3 (4 part.)) | 0
Completed | 0 | 5 (6 participants were re-randomized to track 3 (5 part.) or to track 5 (1 part.)) | 1 | 2 (1 participant was re-randomized to track 5) | 0
Not Completed | 0 | 36 | 15 | 16 | 0
Not completed — Disease progression | 0 | 24 | 13 | 14 | 0
Not completed — Adverse event unrelated to study drug | 0 | 1 | 1 | 1 | 0
Not completed — Study drug toxicity | 0 | 3 | 0 | 1 | 0
Not completed — Participant request to discontinue | 0 | 2 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 3 | 1 | 0 | 0
Not completed — Other reasons | 0 | 3 | 0 | 0 | 0
Period: Track 4
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Started | 0 | 53 | 0 | 60 | 0
Completed | 0 | 2 (1 participant was re-randomized to track 5) | 0 | 18 | 0
Not Completed | 0 | 51 | 0 | 42 | 0
Not completed — Study drug toxicity | 0 | 6 | 0 | 5 | 0
Not completed — Participant request to discontinue | 0 | 1 | 0 | 1 | 0
Not completed — Participant withdrew consent | 0 | 1 | 0 | 0 | 0
Not completed — Other reasons | 0 | 5 | 0 | 3 | 0
Not completed — Disease progression | 0 | 33 | 0 | 32 | 0
Not completed — Adverse event unrelated to study drug | 0 | 5 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Period: Track 5
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Started | 0 | 0 | 0 | 0 | 43 (6 participants had prior treatment in track 1 (1 part.), 2 (2 part.), 3 (2 part.) or 4 (1 part.))
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 43
Not completed — Disease progression | 0 | 0 | 0 | 0 | 34
Not completed — Adverse event unrelated to study drug | 0 | 0 | 0 | 0 | 2
Not completed — Study drug toxicity | 0 | 0 | 0 | 0 | 2
Not completed — Participant request to discontinue | 0 | 0 | 0 | 0 | 3
Not completed — Other reasons | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205 | Total
Number analyzed (Participants) | 49 | 104 | 17 | 88 | 37 | 295
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (10.27) | 63.6 (9.25) | 66.6 (9.17) | 62.3 (9.04) | 63.6 (7.89) | 63.5 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 34 | 8 | 38 | 21 | 122
  Male | 28 | 70 | 9 | 50 | 16 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 5 | 1 | 9
  Not Hispanic or Latino | 25 | 65 | 17 | 58 | 27 | 192
  Unknown or Not Reported | 23 | 37 | 0 | 25 | 9 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 7 | 2 | 2 | 3 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 6 | 1 | 6 | 6 | 19
  White | 42 | 85 | 14 | 78 | 26 | 245
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 0 | 2 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants whose confirmed best overall response (BOR) is either a complete response (CR) or partial response (PR). BOR was assessed by investigator per RECIST1.1.
  Results are presented by study track. Track 1 = participants naive for prior immuno-oncology (IO) therapy and PD-L1 positive Track 2 = participants naive for prior immuno-oncology (IO) therapy and PD-L1 negative Track 3 = participants with prior anti-PD-1/PD-L1 therapy Track 4 = participants naive for prior anti-PD-1/PD-L1 therapy (established upon enrollment closure of tracks 1,2 and 3) Track 5 = participants with prior anti-PD-1/PD-L1 therapy (established upon enrollment closure of tracks 1,2 and 3).
  Results for each study track are presented only for treatment groups who received a treatment in that specific track.
Time Frame: From first dose to 2 years following last dose (up to 30 months)
Population: All treated participants. 14 participants, after receiving initial treatment, were re-randomized to a second, different treatment. They were analyzed under both groups they received treatment for.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Number analyzed (Participants) | 49 | 106 | 18 | 93 | 43
Percent of Participants
  Study Track 1: number analyzed (Participants) | 40 | 4 | 0 | 3 | 0
  Study Track 1 | 17.5 [7.3 to 32.8] | 25.0 [0.6 to 80.6] |  | 0 [0.0 to 70.8] |
  Study Track 2: number analyzed (Participants) | 9 | 8 | 2 | 12 | 0
  Study Track 2 | 0 [0.0 to 33.6] | 0 [0.0 to 33.6] | 0 [0.0 to 84.2] | 25.0 [5.5 to 57.2] |
  Study Track 3: number analyzed (Participants) | 0 | 41 | 16 | 18 | 0
  Study Track 3 |  | 2.4 [0.1 to 12.9] | 0 [0.0 to 20.6] | 5.6 [0.1 to 27.3] |
  Study Track 4: number analyzed (Participants) | 0 | 53 | 0 | 60 | 0
  Study Track 4 |  | 1.9 [0.0 to 10.1] |  | 20.0 [10.8 to 32.3] |
  Study Track 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 43
  Study Track 5 |  |  |  |  | 2.3 [0.1 to 12.3]

2. Primary Outcome: Duration of Response (DOR)
Description: DOR, computed for all treated participants with a confirmed BOR of CR or PR, is defined as the time between the date of first response and the date of first documented disease progression (as determined by RECIST 1.1) or death due to any cause.
  Results are presented by study track. Track 1 = participants naive for prior immuno-oncology (IO) therapy and PD-L1 positive Track 2 = participants naive for prior immuno-oncology (IO) therapy and PD-L1 negative Track 3 = participants with prior anti-PD-1/PD-L1 therapy Track 4 = participants naive for prior anti-PD-1/PD-L1 therapy (established upon enrollment closure of tracks 1,2 and 3) Track 5 = participants with prior anti-PD-1/PD-L1 therapy (established upon enrollment closure of tracks 1,2 and 3).
  Results for each study track are presented only for treatment groups who received a treatment in that specific track.
Time Frame: From first dose to 2 years following last dose (up to 30 months)
Population: All participants with a confirmed best overall response (BOR) of Complete Response (CR) or Partial Response (PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Number analyzed (Participants) | 7 | 3 | 0 | 16 | 1
Months
  Study Track 1: number analyzed (Participants) | 7 | 1 | 0 | 0 | 0
  Study Track 1 | 12.81 [0.0 to NA] — Insufficient number of subjects analyzed | 8.57 [NA to NA] — Insufficient number of subjects analyzed |  |  |
  Study Track 2: number analyzed (Participants) | 0 | 0 | 0 | 3 | 0
  Study Track 2 |  |  |  | NA [NA to NA] — Insufficient number of subjects analyzed |
  Study Track 3: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0
  Study Track 3 |  | NA [NA to NA] — Insufficient number of subjects analyzed |  | NA [NA to NA] — Insufficient number of subjects analyzed |
  Study Track 4: number analyzed (Participants) | 0 | 1 | 0 | 12 | 0
  Study Track 4 |  | NA [NA to NA] — Insufficient number of subjects analyzed |  | 12.65 [8.7 to NA] — Insufficient number of subjects analyzed |
  Study Track 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Study Track 5 |  |  |  |  | 3.75 [NA to NA] — Insufficient number of subjects analyzed

3. Primary Outcome: Progression Free Survival Rate (PFSR) at 24 Weeks
Description: The PFSR at 24 weeks is defined as the proportion of treated participants remaining progression free and surviving at 24 weeks since the first dosing date.
  Results are presented by study track. Track 1 = participants naive for prior immuno-oncology (IO) therapy and PD-L1 positive (>=1%) Track 2 = participants naive for prior immuno-oncology (IO) therapy and PD-L1 negative (<1%) Track 3 = participants with prior anti-PD-1/PD-L1 therapy Track 4 = participants naive for prior anti-PD-1/PD-L1 therapy (established upon enrollment closure of tracks 1,2 and 3) Track 5 = participants with prior anti-PD-1/PD-L1 therapy (established upon enrollment closure of tracks 1,2 and 3).
  Results for each study track are presented only for treatment groups who received a treatment in that specific track.
Time Frame: From first dose to 24 weeks after first dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Number analyzed (Participants) | 49 | 106 | 18 | 93 | 43
Proportion of Participants
  Study Track 1: number analyzed (Participants) | 40 | 4 | 0 | 3 | 0
  Study Track 1 | 0.302 [0.164 to 0.451] | NA [NA to NA] — Insufficient number of participants remaining progression free |  | NA [NA to NA] — Insufficient number of participants remaining progression free |
  Study Track 2: number analyzed (Participants) | 9 | 8 | 2 | 12 | 0
  Study Track 2 | NA [NA to NA] — Insufficient number of participants remaining progression free | NA [NA to NA] — Insufficient number of participants remaining progression free | NA [NA to NA] — Insufficient number of participants remaining progression free | 0.455 [0.167 to 0.707] |
  Study Track 3: number analyzed (Participants) | 0 | 41 | 16 | 18 | 0
  Study Track 3 |  | 0.191 [0.079 to 0.340] | NA [NA to NA] — Insufficient number of participants remaining progression free | NA [NA to NA] — Insufficient number of participants remaining progression free |
  Study Track 4: number analyzed (Participants) | 0 | 53 | 0 | 60 | 0
  Study Track 4 |  | NA [NA to NA] — Insufficient number of participants remaining progression free |  | 0.391 [0.265 to 0.514] |
  Study Track 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 43
  Study Track 5 |  |  |  |  | 0.111 [0.036 to 0.235]

4. Secondary Outcome: Percentage of Participants Experiencing Adverse Events (AEs)
Description: This outcome measure describes the percentage of participants who experienced any grade, all causality AEs during the specified time frame
Time Frame: From first dose to 100 days following last dose
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Number analyzed (Participants) | 49 | 106 | 18 | 93 | 43
Percent of Participants | 100.0 | 100.0 | 100.0 | 98.9 | 100.0

5. Secondary Outcome: Percentage of Participants Experiencing Serious Adverse Events (SAEs)
Description: This outcome measure describes the percentage of participants who experienced any grade, all causality SAEs during the specified time frame
Time Frame: From first dose to 100 days following last dose
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Number analyzed (Participants) | 49 | 106 | 18 | 93 | 43
Percent of Participants | 57.1 | 53.8 | 61.1 | 58.1 | 60.5

6. Secondary Outcome: Percentage of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: This outcome measure describes the percentage of participants who experienced all causality AEs leading to discontinuation of study therapy during the specified time frame
Time Frame: From first dose to 100 days following last dose
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Number analyzed (Participants) | 49 | 106 | 18 | 93 | 43
Percent of Participants | 14.3 | 23.6 | 5.6 | 11.8 | 14.0

7. Secondary Outcome: Percentage of Participants Experiencing Death
Description: This outcome measure describes the percentage of participants who died (due to any cause) during the specified time frame
Time Frame: From first dose to up to 45 months following first dose
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Number analyzed (Participants) | 49 | 106 | 18 | 93 | 43
Percent of Participants | 57.1 | 55.7 | 66.7 | 46.2 | 62.8

8. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities in Hepatic Tests
Description: The following measurements will be considered laboratory abnormalities for hepatic tests:
  * ALT or AST > 3 x ULN, > 5 x ULN, > 10 x ULN and > 20 x ULN
  * Total bilirubin > 2 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN ALT=Alanine aminotransferase AST=Aspartate aminotransferase ULN=Upper Limit of Normal
Time Frame: From first dose to 100 days following last dose (approximately 9 months)
Population: All treated participants with available measurements. 14 participants, after receiving initial treatment, were re-randomized to a second, different treatment. When measurements were available, these participants were analyzed under both groups they received treatment for.
Measure: Number; unit: Participants
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Number analyzed (Participants) | 48 | 97 | 18 | 91 | 43
Participants
  ALT OR AST > 3XULN | 4 | 3 | 1 | 5 | 3
  ALT OR AST > 5XULN | 2 | 0 | 0 | 3 | 2
  ALT OR AST > 10XULN | 2 | 0 | 0 | 1 | 2
  ALT OR AST > 20XULN | 0 | 0 | 0 | 1 | 1
  TOTAL BILIRUBIN > 2XULN | 1 | 0 | 0 | 2 | 3
  Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN | 0 | 0 | 0 | 2 | 2
  Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN | 0 | 0 | 0 | 2 | 2

9. Secondary Outcome: Number of Participants Experiencing Laboratory Abnormalities in Thyroid Tests
Description: The following measurements will be considered laboratory abnormalities for thyroid tests:
  * TSH value > ULN and
  * With baseline TSH value ≤ ULN
  * At least one T3/T4 test value < LLN
  * Low TSH < LLN and
  * With baseline TSH value ≥ LLN
  * At least one T3/T4 test value > ULN TSH = thyroid stimulating hormone ULN=Upper Limit of Normal LLN=Lower Limit of Normal T3=Triiodothyronine T4=Thyroxine
Time Frame: From first dose to 100 days following last dose (approximately 9 months)
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Nivolumab | Nivolumab + Dasatinib | Nivolumab + BMS986016 | Nivolumab + Ipilimumab | Nivolumab + BMS986205
Number analyzed (Participants) | 29 | 76 | 14 | 75 | 35
Participants
  TSH > ULN | 9 | 16 | 3 | 24 | 9
  TSH > ULN WITH TSH <= ULN AT BASELINE | 6 | 9 | 1 | 17 | 6
  TSH > ULN WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN | 4 | 3 | 1 | 8 | 6
  TSH < LLN | 5 | 3 | 0 | 20 | 4
  TSH < LLN WITH TSH >= LLN AT BASELINE | 5 | 1 | 0 | 16 | 4
  TSH < LLN WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN | 3 | 1 | 0 | 5 | 0

ADVERSE EVENTS:
Time Frame: All cause mortality: from first dose to up to 45 months after first dose SAEs and AEs: from first dose to 100 days following last dose
Description: Results are presented by study track. Track 1 = naive for prior immuno-oncology (IO) therapy and PD-L1 positive Track 2 = naive for prior immuno-oncology (IO) therapy and PD-L1 negative Track 3 = with prior anti-PD-1/PD-L1 therapy Track 4 = naive for prior anti-PD-1/PD-L1 therapy (established upon enrollment closure of tracks 1,2 and 3) Track 5 = with prior anti-PD-1/PD-L1 therapy (established upon enrollment closure of tracks 1,2 and 3).
Groups:
- Track 1 - Nivolumab; Track 2 - Nivolumab: Nivolumab monotherapy 240 mg Q2W administered until completion of 6 cycles (1 cycle=4 weeks)
- Track 1 - Nivolumab + Dasatinib; Track 2 - Nivolumab + Dasatinib; Track 3 - Nivolumab + Dasatinib; Track 4 - Nivolumab + Dasatinib: Nivolumab 240 mg Q2W + Dasatinib 100 mg QD, administered until completion of 6 cycles (1 cycle=4 weeks)
- Track 1 - Nivolumab + Ipilimumab; Track 2 - Nivolumab + Ipilimumab; Track 3 - Nivolumab + Ipilimumab; Track 4 - Nivolumab + Ipilimumab: Nivolumab 240 mg Q2W for 12 doses + Ipilimumab 1 mg/kg Q6W for 4 doses, administered until completion of 24 weeks of study
- Track 2 - Nivolumab + BMS986016; Track 3 - Nivolumab + BMS986016: Nivolumab 240 mg Q2W + BMS986016 20 mg Q2W, administered until completion of 6 cycles (1 cycle=4 weeks)
- Track 5 - Nivolumab + BMS986205: Nivolumab 480 mg Q4W + BMS986205 100 mg QD, administered until completion of 6 cycles (1 cycle=4 weeks)
Arm/Group | Track 1 - Nivolumab | Track 1 - Nivolumab + Dasatinib | Track 1 - Nivolumab + Ipilimumab | Track 2 - Nivolumab | Track 2 - Nivolumab + Dasatinib | Track 2 - Nivolumab + BMS986016 | Track 2 - Nivolumab + Ipilimumab | Track 3 - Nivolumab + Dasatinib | Track 3 - Nivolumab + BMS986016 | Track 3 - Nivolumab + Ipilimumab | Track 4 - Nivolumab + Dasatinib | Track 4 - Nivolumab + Ipilimumab | Track 5 - Nivolumab + BMS986205
All-Cause Mortality (participants affected / at risk) | 22/40 | 2/4 | 1/3 | 6/9 | 4/8 | 2/2 | 6/12 | 20/41 | 10/16 | 9/18 | 33/53 | 27/60 | 27/43
Serious Adverse Events (participants affected / at risk) | 24/40 | 2/4 | 0/3 | 4/9 | 5/8 | 2/2 | 5/12 | 17/41 | 9/16 | 10/18 | 33/53 | 39/60 | 26/43
Other Adverse Events (participants affected / at risk) | 38/40 | 4/4 | 3/3 | 9/9 | 7/8 | 2/2 | 12/12 | 38/41 | 16/16 | 17/18 | 50/53 | 59/60 | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Track 1 - Nivolumab (N=40) | Track 1 - Nivolumab + Dasatinib (N=4) | Track 1 - Nivolumab + Ipilimumab (N=3) | Track 2 - Nivolumab (N=9) | Track 2 - Nivolumab + Dasatinib (N=8) | Track 2 - Nivolumab + BMS986016 (N=2) | Track 2 - Nivolumab + Ipilimumab (N=12) | Track 3 - Nivolumab + Dasatinib (N=41) | Track 3 - Nivolumab + BMS986016 (N=16) | Track 3 - Nivolumab + Ipilimumab (N=18) | Track 4 - Nivolumab + Dasatinib (N=53) | Track 4 - Nivolumab + Ipilimumab (N=60) | Track 5 - Nivolumab + BMS986205 (N=43)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Euthanasia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Human chorionic gonadotropin positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 0 | 0 | 2 | 1 | 1 | 1 | 9 | 3 | 3 | 19 | 16 | 13
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brachial plexopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 4 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 3 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Track 1 - Nivolumab (N=40) | Track 1 - Nivolumab + Dasatinib (N=4) | Track 1 - Nivolumab + Ipilimumab (N=3) | Track 2 - Nivolumab (N=9) | Track 2 - Nivolumab + Dasatinib (N=8) | Track 2 - Nivolumab + BMS986016 (N=2) | Track 2 - Nivolumab + Ipilimumab (N=12) | Track 3 - Nivolumab + Dasatinib (N=41) | Track 3 - Nivolumab + BMS986016 (N=16) | Track 3 - Nivolumab + Ipilimumab (N=18) | Track 4 - Nivolumab + Dasatinib (N=53) | Track 4 - Nivolumab + Ipilimumab (N=60) | Track 5 - Nivolumab + BMS986205 (N=43)
Anaemia (Blood and lymphatic system disorders) | 7 | 1 | 0 | 1 | 3 | 0 | 3 | 6 | 2 | 1 | 15 | 10 | 6
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 3 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0
Hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 4 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 6 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 2 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 2 | 5 | 5 | 6 | 6
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 3 | 3 | 0 | 1 | 0 | 3 | 9 | 1 | 2 | 20 | 18 | 13
Diarrhoea (Gastrointestinal disorders) | 13 | 0 | 1 | 2 | 4 | 0 | 4 | 8 | 5 | 2 | 20 | 17 | 11
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 3 | 2 | 3 | 4 | 0 | 3 | 16 | 3 | 4 | 22 | 18 | 16
Oesophageal mucosa erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 3
Tongue dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 1 | 0 | 1 | 3 | 0 | 3 | 8 | 1 | 3 | 14 | 14 | 5
Asthenia (General disorders) | 5 | 2 | 0 | 2 | 1 | 0 | 0 | 4 | 0 | 0 | 11 | 11 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1
Chest pain (General disorders) | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 5 | 3 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 7 | 3 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1
Fatigue (General disorders) | 16 | 1 | 0 | 1 | 4 | 0 | 6 | 19 | 5 | 8 | 27 | 30 | 20
Influenza like illness (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 3 | 2 | 0
Oedema (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 2
Oedema peripheral (General disorders) | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 2 | 7 | 7
Pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 2 | 0
Pyrexia (General disorders) | 3 | 2 | 0 | 1 | 2 | 0 | 2 | 4 | 1 | 3 | 10 | 10 | 5
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 2 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 1 | 2 | 2 | 2
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 4
Urinary tract infection (Infections and infestations) | 7 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 5 | 2 | 5
Amylase increased (Investigations) | 3 | 0 | 1 | 1 | 0 | 1 | 2 | 3 | 0 | 2 | 5 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 1 | 3 | 4 | 4
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 3 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0
Lipase increased (Investigations) | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 2 | 3 | 3 | 2
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 7 | 2 | 1 | 0 | 2 | 0 | 1 | 6 | 0 | 2 | 8 | 11 | 13
Weight increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 16 | 1 | 1 | 2 | 2 | 1 | 1 | 11 | 4 | 5 | 25 | 17 | 15
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 4 | 4
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 4 | 6 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 0 | 2 | 4 | 7 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 1 | 0 | 0 | 1 | 7 | 1 | 2 | 3 | 10 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 0 | 0 | 2 | 4 | 1
Sodium retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 7 | 11 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 2 | 1 | 1 | 1 | 0 | 0 | 8 | 1 | 4 | 6 | 14 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 2 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 3 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | 1 | 1 | 1 | 0 | 1 | 6 | 1 | 2 | 3 | 4 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 3 | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 5 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 0 | 1 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 6 | 2 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 0 | 1 | 1 | 0 | 0 | 2 | 7 | 1 | 3 | 7 | 9 | 3
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 6 | 1 | 2
Headache (Nervous system disorders) | 11 | 0 | 1 | 1 | 3 | 0 | 2 | 5 | 2 | 4 | 8 | 7 | 8
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 1 | 2
Sciatica (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 6 | 0 | 0 | 1 | 2 | 0 | 0 | 4 | 0 | 2 | 9 | 6 | 2
Confusional state (Psychiatric disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 2
Depression (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 5 | 0
Insomnia (Psychiatric disorders) | 7 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 0 | 1 | 5 | 10 | 5
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 1 | 2 | 2 | 0 | 3 | 5 | 2 | 6 | 13 | 15 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 3 | 0 | 2 | 3 | 1 | 1 | 7 | 0 | 6 | 21 | 20 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 4 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 1 | 2 | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 2 | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 10 | 1 | 0 | 7 | 4 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 7 | 5 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 2 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 2 | 2 | 4 | 3
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 1 | 1 | 2 | 1 | 0 | 2 | 4 | 1 | 3 | 5 | 16 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 2 | 0 | 2 | 0 | 0 | 7 | 3 | 3 | 7 | 10 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 6 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 5 | 6
Hypotension (Vascular disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 2 | 2

LIMITATIONS AND CAVEATS:
This study was terminated early by sponsor for reasons unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT02750514/SAP_000.pdf
  • Study Protocol (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02750514/Prot_001.pdf